CLINICAL TRIAL: NCT01954186
Title: When and How to Administer Oxytocin for Active Management of Third Stage of Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etlik Zubeyde Hanim Womens' Health and Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, SEZİN ERTURK AKSAKAL, gynecologist and obstetrician, Etlik Zubeyde Hanim Womens' Health and Teaching Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: EtlikWHTH
Record Dates: First submitted 2013-09-22; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Postpartum Bleeding
Keywords: Oxytocin; Active Management of Third Stage of Labour
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous & intramuscular oxytocin (Experimental): intravenous or intramuscular 10 iu oxytocin
  Interventions: Procedure: after delivery of the fetus & when anterior shoulder seen
- after delivery & when anterior shoulder seen (Active Comparator): oxytocin 10 iu after the delivery of the fetus or when the anterior shoulder was seen after the fetal head was delivered
  Interventions: Drug: intravenous & intramuscular oxytocin

INTERVENTIONS:
Drug: intravenous & intramuscular oxytocin — intravenous or intramuscular 10 iu oxytocin
  Other Names: Postuitrin
  Arms: after delivery & when anterior shoulder seen
Procedure: after delivery of the fetus & when anterior shoulder seen — oxytocin 10 iu after the delivery of the fetus or when the anterior shoulder was seen after the fetal head was delivered
  Arms: intravenous & intramuscular oxytocin

SUMMARY:
To compare the efficacy of the route and timing of oxytocin administration for Active management of third stage of labour (AMTSL).

DETAILED DESCRIPTION:
Our objective is to determine the most efficient route and timing of oxytocin administration by measuring the duration of third stage of labour, quantitative blood during the first hour after delivery and comparing haemoglobin and haematocrit changes and the need for additional interventions in patients who had either a spontaneous labour or received labour augmentation with oxytocin.

ELIGIBILITY:
Inclusion Criteria:

* having a singleton pregnancy above 37th gestational week
* normal live vaginal delivery with cephalic presentation
* being in active labor

Exclusion Criteria:

* Fetal demise
* multiple pregnancy
* known coagulation disorder
* presentation anomalies
* placental pathology
* liver disease
* thrombocytopenia
* hypertension or being currently on anticoagulants
* having a cesarean section, operative delivery or deep vaginal tear
* chorioamnionitis
* developing HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count) or DIC (disseminated intravascular coagulation) before delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
postpartum bleeding in the third stage of labour | participants will be followed for the duration of hospital stay, an expected average of 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Berna DILBAZ, Assoc. Prof., Study Director — Etlik Zübeyde Hanım Women's Health Teaching and Research Hospital, Obstetrics and Gynecology, Ankara, Turkey ,; Emire OGUZ ORHAN, MD, Study Chair — Sivas State Hospital; Sezin ERTURK AKSAKAL, MD, Principal Investigator — Etlik Zübeyde Hanım Women's Health Teaching and Research Hospital, Obstetrics and Gynecology, Ankara, Turkey; Sibel ALTINBAS, Assist. Prof., Study Chair — Hacettepe University Kastamonu Medical Faculty, Obstetrics and Gynecology, Ankara, Turkey,; Salim ERKAYA, Assoc. Prof., Study Chair — Zekai Tahir Burak Maternity and Teaching Hospital, Obstetrics and Gynecology, Ankara, Turkey
Locations (1):
- Etlik Zübeyde Hanım Women's Health Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Oladapo OT, Okusanya BO, Abalos E, Gallos ID, Papadopoulou A. Intravenous versus intramuscular prophylactic oxytocin for the third stage of labour. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD009332. doi: 10.1002/14651858.CD009332.pub4. PMID 33169839
- [Derived] Oguz Orhan E, Dilbaz B, Aksakal SE, Altinbas S, Erkaya S. Prospective randomized trial of oxytocin administration for active management of the third stage of labor. Int J Gynaecol Obstet. 2014 Nov;127(2):175-9. doi: 10.1016/j.ijgo.2014.05.022. Epub 2014 Jul 17. PMID 25108586